CLINICAL TRIAL: NCT01431703
Title: The Learning Curve of NBI With Magnification in the Diagnosis of Colorectal Lesions
Status: Completed | Type: Observational
Sponsor: Zhizheng Ge (Other)
Responsible Party: Sponsor-Investigator, Zhizheng Ge, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: rjyyxhk0923
Record Dates: First submitted 2011-09-08; First posted 2011-09-09 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Colorectal Lesion
Keywords: narrow band imaging; learning curve; colorectal; differential diagnosis; with colorectal lesion; NBI with magnification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — if the lesion is neoplastic or sm deeper cancer, we just take biopsy.If the lesion is adenomatous or sm1-2 cancer,we do polypectomy, EMR or ESD to get the specimen.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It exists a learning curve in using NBI with magnification to differentiating colorectal lesions.

DETAILED DESCRIPTION:
It is very useful to use narrow-band imaging and Sano CP analysis in the differential diagnosis of colorectal lesions. The endoscopists who had never used NBI or no knowledge of NBI can have effective and stable diagnostic accuracy after using NBI with magnification to diagnose 15 target and non-target lesions respectively.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16 to 85
* Any patient undergoing NBI with magnification colonoscopy exam and found with colorectal lesions

Exclusion Criteria:

* Unwilling to consent
* Had surgery of colorectal tumors
* Using NSAIDS
* Diagnosed or suspected IBD
* Familial adenomatous polyposis(FAP) or hereditary non-polyposis colorectal(HNPCC) or other hereditary disease

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: academic hospital endoscopist of digestive department
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NBI With Magnification: Patients with lesions diagnosed by Sano classification using NBI with magnification
Period: Overall Study
Arm/Group | NBI With Magnification
Started | 326
Completed | 326
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NBI With Magnification
Number analyzed (Participants) | 326
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 229
  >=65 years | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.9)
Gender [Count of Participants; unit: Participants]
  Female | 131
  Male | 195
Region of Enrollment [Number; unit: participants]
  China | 326

OUTCOME MEASURES:

1. Primary Outcome: Accuracy, Sensitivity, and Specificity for Differentiating Neoplastic and Non-neoplastic Lesions
Time Frame: For this training, patients were consecutively enrolled until a total of 45 target and non-target lesions were obtained.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Arm/Group | NBI With Magnification
Number analyzed (Participants) | 326
percentage of lesions
  Accuracy | 94.3 [91.5 to 97.1]
  Sensitivity | 98.0 [94.3 to 99.9]
  Specificity | 92.0 [88.5 to 95.6]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | NBI With Magnification
Serious Adverse Events (participants affected / at risk) | 0/326
Other Adverse Events (participants affected / at risk) | 0/326

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No